CLINICAL TRIAL: NCT06553547
Title: 4-Week, Multi-Center, Randomized, Db-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Safety & Efficacy of Tenapanor for the T/t of IBS-C in Pts. 6 to < 12 Yrs. Old
Brief Title: 4-Week, Multi-center Dose-Ranging Study for the IBS-C in Pts. 6 to <12 Yrs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEN-01-202
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)
Keywords: IBS-C
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Tenapanor Cohort 1 (Experimental): Tenapanor 2 mg BID
  Interventions: Drug: Tenapanor
- Tenapanor Cohort 2 (Experimental): Tenapanor 5 mg BID
  Interventions: Drug: Tenapanor
- Tenapanor Cohort 3 (Experimental): Tenapanor 10 mg BID
  Interventions: Drug: Tenapanor
- Tenapanor Cohort 4 (Experimental): Tenapanor 15 mg BID
  Interventions: Drug: Tenapanor
- Tenapanor Cohort 5 (Experimental): Tenapanor 20 mg BID
  Interventions: Drug: Tenapanor
- Tenapanor Cohort 6 (Experimental): Tenapanor 25 mg BID
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor — Tenapanor 5 mg/mL solution
  Other Names: IBSRELA
  Arms: Tenapanor Cohort 1; Tenapanor Cohort 2; Tenapanor Cohort 3; Tenapanor Cohort 4; Tenapanor Cohort 5; Tenapanor Cohort 6
Drug: Placebo — Matching Placebo solution
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled dose-ranging study to assess the safety and efficacy of tenapanor for treatment of the IBS-C in pediatric patients 6 to less than 12 year old.

DETAILED DESCRIPTION:
This study consists of 2 week screening period in which subjects who have consented will be evaluated for eligibility per protocol requirements. During this 2 week screening period subjects will be given access to ediary in which they will be required to self report symptoms of IBS-C daily. Information in ediary will also be used to determine eligibility prior to enrollment.

During the 4 week RTP (Randomized treatment period), subjects will be randomized in in a ratio of 5:1 to receive tenapanor or matching placebo for 4 weeks. During the RTP, patients will continue recording daily assessments in the eDiary system as instructed and compliance with eDiary entries will be monitored. Patients will return for study visit every weeks (Visits 3-6) and will undergo safety assessments as per the protocol. At the end of this 4 week period, subjects will complete 2 week treatment free follow-up period and safety assessments per protocol will be conducted at the end of this 2 week period.

The study plans to enroll up to 6 cohorts of eligible patients sequentially, starting from Cohort 1 with 12 patients randomized in to receive tenapanor 2 mg BID or matching placebo for 4 weeks. Subsequent cohorts will assess increasing tenapanor doses, following a dose escalation order. The study will proceed to the next dosing cohort if the current cohort completes the 4-week RTP and does not meet any of the dose escalation stopping criteria pre-specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. ≥6 and <12 years old at the Screening visit (Visit 1)
2. Confirmation of negative pregnancy test and use of appropriate contraceptive (including abstinence) in female subjects that have experienced menarche and are of child-bearing potential.
3. Meet the Modified Diagnostic Rome IV criteria for child/adolescent diagnosis of IBS-C
4. Patient is willing to discontinue any laxatives used in favor of the protocol-permitted rescue medicine (which will only be allowed after 72 hours with no bowel movement)
5. Meet the entry criteria assessed during the 2-week Screening period
6. Ability of both the patient and parent/guardian/LAR to communicate with the Investigator and to comply with the requirements of the entire study, including an understanding of the assessments in the eDiary and how to use the eDiary device
7. Patient must provide verbal assent and the parent/guardian/LAR must provide written informed consent before the initiation of any study-specific procedures

Exclusion Criteria:

1. Functional diarrhea as defined by Modified Rome IV child/adolescent criteria
2. IBS with diarrhea (IBS-D), mixed IBS (IBS-M), or unsubtyped IBS as defined by Modified Rome IV child/adolescent criteria
3. History of non-retentive fecal incontinence;
4. Required manual disimpaction any time prior to randomization (after consent)
5. Currently has both unexplained and clinically significant alarm symptoms (lower gastrointestinal [GI] bleeding [rectal bleeding or heme-positive stool], iron-deficiency anemia, or any unexplained anemia, or weight loss) and systemic signs of infection or colitis, or any neoplastic process.
6. Patient has any of the following conditions:

   1. Celiac disease, or positive serological test for celiac disease and the condition has not been ruled out by endoscopic biopsy;
   2. Cystic fibrosis;
   3. Hypothyroidism that is untreated or treated with thyroid hormone at a dose that has not been stable for at least 3 months prior to the Screening Visit;
   4. Down's syndrome or any other chromosomal disorder;
   5. Active anal fissure (Note: History of anal fissure is not an exclusion);
   6. Anatomic malformations (eg, imperforate anus, anal stenosis, anterior displaced anus);
   7. Intestinal nerve or muscle disorders (eg, Hirschprung disease, visceral myopathies, visceral neuropathies);
   8. Neuropathic conditions (eg, spinal cord abnormalities, neurofibromatosis, tethered cord, spinal cord trauma);
   9. Lead toxicity, hypercalcemia;
   10. Neurodevelopmental disabilities
   11. Inflammatory bowel disease
   12. Childhood functional abdominal pain syndrome
   13. Childhood functional abdominal pain
   14. Poorly treated or poorly controlled psychiatric disorders that might influence his or her ability to participate in the study;
   15. Lactose intolerance that is associated with abdominal pain or discomfort and could confound the assessments in this study
   16. History of cancer other than treated basal cell carcinoma of the skin;
   17. History of diabetic neuropathy.
7. Use of medications that are known to affect stool consistency (Prohibited Medications), including fiber supplements, anti-diarrheals, cathartics, antacids, opiates, prokinetic drugs, laxatives, enemas, antibiotics during the Screening period; unless specified as rescue medication, and used accordingly as directed by the Investigator.
8. Patient has had surgery that meets any of the following criteria:

   1. Surgery to remove a segment of the GI tract at any time before the Screening Visit;
   2. Surgery of the abdomen, pelvis, or retroperitoneal structures during the 6 months before the Screening Visit;
   3. An appendectomy or cholecystectomy during the 60 days before the Screening Visit;
   4. Other major surgery during the 30 days before the Screening Visit
9. History of alcohol or substance abuse
10. Participation in other clinical trials within 1 month prior to Screening
11. Patient and/or parent/guardian/LAR is involved in the conduct and/or administration of this trial as an investigator, sub-investigator, trial coordinator, or other staff member, or the patient is a first-degree family member, significant other, or relative residing with one of the above persons involved in the trial
12. If, in the opinion of the Investigator, the patient is unable or unwilling to fulfill the requirements of the protocol or has a condition, which would render the results uninterpretable

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Average weekly SBM (week 4) | 4 weeks
  Change from baseline in average weekly SBM frequency in Week 4

SECONDARY OUTCOMES:
Average weekly SBM (weeks 1, 2 and 3) | 3 weeks
  Change from baseline in average weekly SBM frequency in Week 1, Week 2, and Week 3
SBM Response | 6 weeks
  Weekly ≥3 SBM response: achieving an average weekly SBM frequency ≥3 for a given week
Stool consistency | 6 weeks
  Percent change from baseline in average weekly stool consistency score in each week
  Scale Range:
  1. one (1)= Rabbit droppings: separate hard lumps, like nuts (hard to pass)
  2. seven (7) for Gravy: watery, no solids pieces, entirely liquid"
Abdominal Pain Score | 6 weeks
  Percent change from baseline in average weekly abdominal pain score in each week
  Scale Range:
  zero (0) = no pain and ten (10)= very severe abdominal pain
Rescue medication | 6 weeks
  Overall use of rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Susan Edelstein, PhD, Study Director — Ardelyx
Locations (17):
- United States (17):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Waterway Research & Associates Corp., Miami, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Orlando Health, Inc.- APH Center for Digestive Health and Nutrition, Orlando, Florida
  - Florida Pharmaceutical Research and Associates, Inc., South Miami, Florida
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Mankato Clinic Children's Health Center, Mankato, Minnesota
  - Boys Town National Research Hospital, Boys Town, Nebraska
  - One Perkins Square, Akron, Ohio
  - Prisma Health Children's Hospital, Greenville, South Carolina
  - Maspons Pediatric Gastro, El Paso, Texas
  - Proactive El Paso, LLC, El Paso, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - Pioneer Research Solutions Inc, Sugar Land, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia
  - University Physicians and Surgeons, Inc, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No